CLINICAL TRIAL: NCT03791736
Title: Evaluation of Impact of Sandostatin® Injection Before Axillary Clearance on Lymphocele Formation In Patients With Breast Cancer
Brief Title: Evaluation of Impact of Sandostatin® Injection Before Axillary Clearance on Lymphocele Formation
Acronym: SANDOSTATINE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The surgical technique is no longer used
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015-03
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer; Lymphocele
Keywords: breast cancer; axillary clearance; lymphocele
MeSH Terms: conditions — Breast Neoplasms; Lymphocele | interventions — Octreotide

STUDY DESIGN:
Intervention Model Description: A phase II prospective, single-center, non-randomized study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sandostatine (Experimental): Injection of Sandostatine
  Interventions: Procedure: Injection of sandostatine

INTERVENTIONS:
Procedure: Injection of sandostatine — Intramuscular injection of sandostatin 30 mg 3 days before surgery
  Other Names: Octreotide

SUMMARY:
The lymphocele is the main early postoperative complication of axillary clearance for breast cancer patients with rates up to 85%.

The usual treatment consists of external drainage. However, this method increases the duration of hospitalization.

As a result, some practitioners have abandoned drainage, allowing for ambulatory surgery.

If this solution makes it possible to reduce the duration of the hospitalizations, it involves iterative punctures of the axillary hollow in case of lymphocele These punctures may be responsible for pain, hematoma or infection of the operative site.

To date, no method has proved superior in terms of decreasing the incidence of lymphocele postoperatively axillary clearance.

Octreotide (Sandostatin®) is a peptide, one of whose effects is to reduce the inflammation responsible for lymphoceles.

The aim of the study is to inject Sandostatin® before surgery, with the aim of reducing the incidence of seroma by 50% after axillary clearance

ELIGIBILITY:
Inclusion Criteria:

Breast cancer, histologically proven Axillary clearance Elective axillary approach Age ≥ 18 years OMS < 3 Normal hematological and hepatic blood tests Obtaining the signed written consent of the patient

Exclusion Criteria:

Axillary clearance with a mastectomy Metastatic disease Disorder precluding understanding of trial information or informed consent Pregnancy, breastfeeding women Patient is willing and able to comply with the protocol for the duration of the study including all scheduled treatment, visits and examinations No severe or uncontrolled diabetes Known hypersensitivity to Octreotide Patient with vitamin B12 deficiency Anticoagulant treatment History of cardiovascular disease Other product being tested in the 4 weeks prior to the start of treatment Patient has valid health insurance

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-06 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
A 50% decrease in the incidence of lymphocele (30% to 15% progression) following axillary clearance of patients operated for breast cancer (excluding mastectomy) pretreated with an injection of Sandostatin®. | 6 months
  The frequency of occurrence of a lymphocele requiring at least one evacuation puncture.

SECONDARY OUTCOMES:
Evaluation of the volume of the punctures | 6 months
  Determined by the volume of the punctures carried out
Evaluation of the cost of this treatment | 6 months
  Determined by the data recovered from the Health Insurance

CONTACTS AND LOCATIONS:
Overall Officials: EMMANUELLE MARTIN, MD, Study Director — INSTITUT DE CANCEROLOGIE DE L'OUEST

IPD SHARING:
Plan to Share IPD: No